CLINICAL TRIAL: NCT00475774
Title: The Effect of Body Fat Distribution on the Physiological Response to a Dietary Fat Intervention
Brief Title: Body Fat Distribution and Fat Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TNO (Other)
Collaborators: Netherlands: Ministry of Health, Welfare and Sports (Other Government)
Responsible Party: Dr. W.J. Pasman, TNO Quality of Life
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: P7261
Record Dates: First submitted 2007-05-18; First posted 2007-05-21 (Estimated); Last update posted 2008-04-07 (Estimated); Status verified 2008-04

CONDITIONS: Obesity; Metabolic Disease
MeSH Terms: conditions — Obesity; Metabolic Diseases | interventions — Neprilysin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Long-chain (C18:2) and medium chain fatty acid (C8 and C10).

SUMMARY:
The primary purpose of the study is to examine the effect of body fat distribution on the physiological response to a dietary fat intervention. Physiological response will be evaluated as fatty acid kinetics (plasma and subcutaneous fat appearance).

Secondary objectives are targeted protein production (apoB and adiponectin). Examination of the effect of chain length of the dietary fatty acids on fat tissue characteristics and the effect of chain length on satiety, will be studied as well.

DETAILED DESCRIPTION:
Rationale: The increased prevalence of obesity and the related risk for metabolic diseases have resulted in increased interest in prevention of obesity through life-style interventions. The site of fat storage (visceral or subcutaneous) is considered to be relevant in terms of risk for metabolic disorders. The type of fat consumed may determine storage in either fat storage site and hence be related to metabolic disorders. Long-chain fatty acids have been suggested to be preferentially targeted to subcutaneous fat, whereas medium chain fatty acids may preferably be targeted to the visceral fat depot.

Objective: The primary objective is to examine the effect of body fat distribution on the physiological response to a dietary fat intervention. Physiological response will be evaluated as fatty acid kinetics (plasma and subcutaneous fat appearance), targeted protein production (apoB and adiponectin) and satiety.

Study design: The study is designed as a randomized, double-blind, cross-over trial. Two treatments will be supplied for three weeks, with a wash-out period of at least 3 weeks in-between.

Study population: Twelve apparently healthy overweight/obese men (30-60 years of age) with a BMI of 27-35 kg.m-2 (6 upper body obese (high WHR) en 6 lower body obese (low WHR)).

Intervention: Three weeks intervention with a fat replacement containing long chain fatty acids and three weeks intervention with a fat replacement containing medium chain fatty acids. The margarines will replace the normally consumed margarine. Consumption will take place with breakfast, lunch and dinner.

Main study parameters/endpoints: On the last day of each treatment period subjects will come to TNO for evaluation of the effect of the dietary intervention on fat metabolism and fat tissue. This will be examined with stable isotope techniques and fat biopsies of subcutaneous fat. At baseline subjects will have a total body scan in the MRI to characterize body fat.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Males aged between 30 - 60 years at Day 01 of the study
* Body Mass Index (BMI) between 27-35 kg/m2
* Range in waist-hip ratio as high as possible (preferably <0.90 or >0.95)
* Regular Dutch eating habits and used to consume margarine;
* Non restrained eater
* Voluntary participation
* Having given written informed consent
* Willing to comply with the study procedures
* Agree to be informed about chance findings of pathology found with the MRI
* Willing to accept use of all nameless data, including publication, and the confidential use and storage of all data for at least 15 years
* Willing to accept the disclosure of the financial benefit of participation in the study to the authorities concerned.

Exclusion Criteria:

* Participation in any clinical trial including blood sampling and/or administration of substances up to 90 days before Day 01 of this study
* Having a history of medical or surgical events that may significantly affect the study outcome
* Use of medication that may influence appetite, and/or sensory functioning
* Smoking
* Alcohol consumption (> 28 units/week)
* Contra-indication to MRI scanning
* Reported unexplained weight loss or gain of > 2 kg in the month prior to the pre-study screening
* Reported slimming or medically prescribed diet
* Reported vegan, vegetarian or macrobiotic
* Recent blood donation (<1 month prior to the start of the study)
* Not willing to give up blood donation during the study
* Not having a general practitioner
* Not willing to accept information-transfer concerning participation in the study, or information regarding his health to and from his general practitioner.

Ages: 30 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2007-05; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
fatty acid kinetics (in plasma and subcutaneous fat) | 3 weeks
lipoprotein and adiponectin metabolism | 3 weeks

SECONDARY OUTCOMES:
visual analogue scales to evaluate satiety | 3 weeks
body weight | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Wilrike Pasman, PhD, Principal Investigator — TNO
Locations (1):
- TNO Quality of Life, Zeist, Netherlands